

#### FINAL STATISTICAL ANALYSIS PLAN

### ALKS 3831-A308 NCT03201757

Study Title: A Phase 3 Study to Assess the Long Term Safety, Tolerability and

Durability of Treatment Effect of ALKS 3831 in Subjects with Schizophrenia, Schizophreniform Disorder, or Bipolar I Disorder

Document Status: Version 1.0

Document Date: 13 Jun 2023

Based on: ALKS 3831-A308 Protocol Amendment 3.0 Date: 09 May 2019 and

ALKS 3831-A308 Interim Statistical Analysis Plan 1.0 Date:

06 Jun 2019

Sponsor: Alkermes, Inc.

852 Winter Street Waltham, MA 02451

USA

#### CONFIDENTIAL

Information and data in this document contain trade secrets and privileged or confidential information, which is the property of Alkermes, Inc. No person is authorized to make it public without the written permission of Alkermes, Inc. These restrictions or disclosures will apply equally to all future information supplied to you that is indicated as privileged or confidential. This study is being conducted in compliance with good clinical practice, including the archiving of essential documents.

# TABLE OF CONTENTS

| TABLE ( | OF CONTENTS | 2 |
|---|---|---|
| LIST OF | TABLES | 3 |
| LIST OF | FIGURES | 4 |
| ABBREV | VIATIONS | 5 |
| 1. | INTRODUCTION | 6 |
| 1.1. | Study Objectives | 6 |
| 1.1.1. | Primary Objective | 6 |
| 1.2. | Summary of the Study Design | 6 |
| 2. | SAMPLE SIZE CONSIDERATION | 7 |
| 3. | DATA ANALYSIS | 7 |
| 3.1. | General Statistical Methodology | 7 |
| 3.2. | Definitions of Analysis Populations | 7 |
| 3.2.1. | Safety Population | 7 |
| 3.2.2. | Follow-up Safety Population | 8 |
| 3.2.3. | Post-discontinuation Safety Population | 8 |
| 3.3. | Disposition | 9 |
| 3.4. | Demographics and Baseline Characteristics | 9 |
| 3.5. | Prior and Concomitant Medication | 9 |
| 3.6. | Treatment Adherence Rate and Extent of Exposure to Study Drug | 9 |
| 3.6.1. | Treatment Adherence Rate | 9 |
| 3.6.2. | Extent of Exposure to Study Drug | 9 |
| 3.7. | Efficacy Analyses | 10 |
| 3.7.1. | Efficacy Analysis | 10 |
| 3.7.2. | Multiple Comparison / Multiplicity | 11 |
| 3.7.3. | Subgroup Analysis | 11 |
| 3.7.4. | Other Endpoints | 12 |
| 3.8. | Safety Analysis | 12 |
| 3.8.1. | Adverse Events | 12 |
| 3.8.1.1. | Deaths, Serious and Other Significant AEs | 13 |
| 3.8.1.2. | AEs of Special Interest | 13 |
| 3.8.2. | Clinical Laboratory Parameters | 13 |

| 3.8.3. | Vital Signs and Body Weight | 16 |
|---|---|---|
| 3.8.3.1. | Vital Signs | 16 |
| 3.8.3.2. | Weight and Body Mass Index | 17 |
| 3.8.4. | Columbia-Suicide Severity Rating Scale (C-SSRS) | 17 |
| 3.9. | Pharmacokinetic/ Pharmacodynamic Data Analysis | 18 |
| 4. | INTERIM ANALYSES | 18 |
| 5. | CHANGES IN CONDUCT OR PLANNED ANALYSES FROM THE PROTOCOL | 18 |
| 6. | DEFINITIONS AND CONVENTIONS FOR HANDLING OF THE DATA | |
| 6.1. | Analysis Visit Windows | 19 |
| 6.2. | Handling of Partial Dates of Concomitant Medication and Adverse Events | 21 |
| 6.3. | Handling of Safety Data | 21 |
| 7. | GENERAL STATISTICAL METHODOLOGY (AND REPORTING OF RESULTS) | 22 |
| 7.1. | Reporting Precision | 22 |
| 8. | PROGRAMMING SPECIFICATIONS | 22 |
| 9. | MOCK TABLES, LISTINGS AND FIGURES (TLFS) | 22 |
| 10. | REFERENCES | 23 |
| APPEND | IX 1. AESI - MOVEMENT DISORDERS (INCLUDING<br>EXTRAPYRAMIDAL SYNDROME AND TARDIVE DYSKINESIA;<br>STANDARDIZED MEDDRA QUERY) | 24 |
| APPEND | IX 2. AESI - SUICIDAL IDEATION AND BEHAVIOR (CUSTOM MEDDRA QUERY) | 28 |
| APPEND | IX 3. AE TERMS - ABUSE POTENTIAL (CUSTOM MEDDRA QUERY) | 29 |
| APPEND | IX 4. AE TERMS – DEPENDENCE (CUSTOM MEDDRA QUERY) | 32 |
| APPEND | IX 5. AE TERMS – WITHDRAWAL (CUSTOM MEDDRA QUERY) | 33 |
| APPEND: | IX 6. COVID-19 ANALYSIS | 35 |
| | LIST OF TABLES | |
| Table 1: | Definition of Shift CGI-S Categories | 10 |
| Table 2: | Shift Categories for CGI-S response | 11 |
| Table 3: | Criteria of Potentially Clinically Significant (PCS) Abnormality for Selected Analytes | 14 |

| Table 4: | Shifts Category from Baseline to Any Postbaseline for Selected Lipid | |
|---|---|---|
| | Parameters | 15 |
| Table 5: | Shift Category from Baseline to Any Postbaseline in Glucose and HbA1c | 16 |
| Table 6: | Shift Category from Baseline to Any Postbaseline in Liver Function Test | 16 |
| Table 7: | Criteria for Potentially Clinically Significant (PCS) Blood Pressure or Pulse Rate | 17 |
| Table 8: | Criteria for Potentially Clinically Significant (PCS) Changes from Baseline in Body Weight | 17 |
| Table 9: | C-SSRS Categories for Analysis | 18 |
| Table 10: | Visit Window Definition for Weight, Waist Circumference and CGI-S Data | 19 |
| Table 11: | Visit Window Definition for Vital Signs, Lab and IWQOL-Lite Data | 21 |
| Table 12: | Degree of Precision. | 22 |
| | LIST OF FIGURES | |
| Figure 1: S | Study Design Schematic | 7 |

# **ABBREVIATIONS**

| Abbreviation or Term | Explanation or Definition |
|----------------------|----------------------------------------------|
| AE | Adverse event |
| BMI | Body mass index |
| CGI-S | Clinical Global Impression - Severity |
| CI | Confidence interval |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| CMQ | Customized MedDRA queries |
| eCRF | Electronic case report form |
| EPS | Extra pyramidal symptoms |
| HbA1C | Hemoglobin A1c |
| SAP | statistical analysis plan |
| IWQOL | Impact of Weight on Quality of Life |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NDA | New Drug Application |
| OLZ | Olanzapine |
| PCS | Potentially clinically significant |
| PK | Pharmacokinetic |
| PT | Preferred term |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SMQ | Standardized MedDRA queries |
| SOC | System organ class |
| TEAE | Treatment-emergent adverse event |
| ULN | Upper limit of normal |
| WHO | World Health Organization |

#### 1. INTRODUCTION

This statistical analysis plan (SAP) describes the statistical methods to be used for analyses and presentation of safety and efficacy data for study ALK3831-A308 to support the clinical study report (CSR) development. This document has been prepared based on Alkermes ALKS 3831-A308 Study Protocol Amendment 3.0 (dated 09 May 2019) and Alkermes ALKS 3831-A308 Interim Statistical Analysis Plan to Support New Drug Application (NDA) Submission (dated 09 Jun 2019).

Subjects who have completed or prematurely discontinued ALKS 3831 will be included in the analysis described in this document.

### 1.1. Study Objectives

#### 1.1.1. Primary Objective

The primary objective of this study is to evaluate the long-term safety, tolerability, and durability of treatment effect of ALKS 3831 in subjects with schizophrenia, schizophreniform disorder, or bipolar I disorder.

#### 1.2. Summary of the Study Design

Subjects are eligible to be enrolled in the study within 7 days after completing the antecedent studies (ALK3831-A304, ALK3831-A306, or ALK3831-A307).

Subjects enrolled in the study will be started on the same olanzapine dose that they had maintained at the end of the antecedent study. Available doses of ALKS 3831 will be 5, 10, 15, and 20 mg olanzapine combined with 10 mg samidorphan (henceforth to be referred to as 5/10, 10/10, 15/10, and 20/10 mg). Subjects may be titrated to a different dose after the start of the study at the Investigator's discretion. Dosing will be flexible throughout the study; however, frequent adjustments are discouraged. Dose adjustments will only be performed on-site at the study center. Subjects requiring dose adjustments between scheduled visits will need to arrange an unscheduled visit.

Safety assessments will include adverse event (AE) monitoring, clinical laboratory testing, vital signs, body weight and the Columbia-Suicide Severity Rating Scale (C-SSRS). Psychiatric symptoms will be evaluated using the Clinical Global Impressions-Severity (CGI-S) scale. Additional assessments will include Impact of Weight on Quality of Life-Lite Questionnaire (IWQOL-Lite).

A schematic of the study design is provided in Figure 1.

**Figure 1: Study Design Schematic** 



<sup>a</sup>Visits will occur monthly throughout the 48-month Treatment period. Subjects will start the study on the equivalent olanzapine dose to what they maintained at the end of the antecedent study. The dose may be adjusted to either 5/10, 10/10, 15/10, or 20/10mg throughout the study period based on investigator discretion, and such dose adjustments will require subjects to visit the study site.

#### 2. SAMPLE SIZE CONSIDERATION

No formal sample size calculation is performed for this extension study. A sample size of approximately 500 is based on the estimated maximum number of subjects who might be expected to continue from the antecedent Phase 3 studies within 7 days (ALK3831-A304, ALK3831-A306, or ALK3831-A307).

#### 3. DATA ANALYSIS

### 3.1. General Statistical Methodology

Baseline for efficacy or safety analyses is defined as the last non-missing assessment before the first dose of ALKS 3831 in the ALK3831-A308 study, and it will be used for all efficacy and safety analyses, unless specified otherwise.

All results from this analysis will be presented for the overall group, ie all subjects as a single group, and not by previous treatment sequence in antecedent studies of ALK3831-A303 and ALK3831-A305.

In general, descriptive statistics: n, mean, standard deviation (SD), median, minimum, and maximum, for continuous variables and number and percentage of subjects in each category for categorical variables will be provided.

All source data will be presented as subject data listings.

# 3.2. Definitions of Analysis Populations

#### 3.2.1. Safety Population

The Safety Population will include all subjects who enrolled and received at least one dose of ALKS 3831 in the ALK3831-A308 study. All analyses will be conducted using the Safety Population except for AEs in the safety follow-up period and AE to evaluate the potential for

drug withdrawal and dependence. The populations used for the analyses of these events are specified below.

#### **3.2.2.** Follow-up Safety Population

Follow-up Safety Population will be defined as subjects in the Safety Population and met any of the following criteria:

- Completed at least one follow-up visit after >7 days of the last dose of ALKS 3831
- Reported at least one AE after >7 days of the last dose of ALKS 3831
- Follow-up Safety Population will be used to analyze the AEs in the safety follow-up period

#### 3.2.3. Post-discontinuation Safety Population

Post-discontinuation Safety Population will be defined as subjects in the Safety Population and met any of the following criteria:

- Completed at least one follow-up visit >2 days after the last dose of ALKS 3831
- Reported at least one AE >2 days after the last dose of ALKS 3831

AEs to evaluate potential for drug withdrawal and dependence emerging following discontinuation of ALKS 3831 will be assessed for this population, during the period of >2 days to 16 days after the last dose of drug for subjects with at least 4 weeks ALKS 3831 exposure.

#### 3.3. Disposition

The number and percentage of subjects completing or prematurely discontinuing the study including reasons for discontinuation will be summarized for the following:

- Subjects who enrolled in the study
- Subjects in the Safety Population
- Subjects who completed the treatment period
- Subjects who discontinued treatment along with reason for discontinuation
- Subjects who are ongoing in the treatment period

### 3.4. Demographics and Baseline Characteristics

Demographics and baseline characteristics such as sex, age, race, ethnicity, weight, and body mass index (BMI) will be summarized for the Safety Population.

#### 3.5. Prior and Concomitant Medication

Prior medications will be defined as medications taken prior to the first dose of study drug in ALK3831-A308 study. Concomitant medications will be defined as medications taken on or after the first dose of study drug in ALK3831-A308 study. All medications will be coded using the World Health Organization WHO-DD Enhanced + Herbal (version: March 2016).

Concomitant medications taken during the treatment period will be summarized by the preferred name, for the Safety Population. All reported medications (including those initiated after the last dose of study medication) will be included in the listing. For the summary table, if a subject has taken a concomitant medication more than once, the subject will be counted only once for that medication.

## 3.6. Treatment Adherence Rate and Extent of Exposure to Study Drug

#### 3.6.1. Treatment Adherence Rate

Treatment adherence to the daily dosing schedule during treatment period will be summarized. Treatment adherence will be calculated as follows:

$$100 \times \frac{\text{Total tablets dispensed} - \text{total tablets returned} - \text{total tablets lost}}{\text{Total tablets scheduled to be taken}}$$

#### 3.6.2. Extent of Exposure to Study Drug

Duration of exposure to study drug (ALKS 3831) is defined as the number of days from the date of the first dose of study drug in this study (ALK3831-A308) to the date of the last dose of study drug, inclusive (ie, last dose date – first dose date + 1 day). Duration of exposure to study drug will be summarized for the Safety Population.

The overall mean and modal dose of olanzapine will be summarized. Number and percentage of subjects will be summarized by their modal dose level and final dose level. Summary of the

extent of exposure will also be presented by demographic subgroups: Age, Sex, Race, Region, weight, and body mass index (BMI). Dose level will be summarized by visit at 12 months, 18 months, 24 months, and 48 months.

Dose level at 12 months, 18 months 24 months, and 48 months will be summarized by antecedent study.

#### 3.7. Efficacy Analyses

#### 3.7.1. Efficacy Analysis

The following efficacy endpoints will be analyzed:

- Change from baseline in CGI-S score by visit
- Shift analysis in CGI-S
- Change from baseline in IWQOL-Lite scales (total score, physical function, self-esteem, sexual life, public distress, and work) by visit
- Time to treatment discontinuation

Value and change from baseline in CGI-S and IWQOL-Lite scores by visit will be summarized using descriptive statistics.

The IWQOL-Lite scale is a 31-item self-report measure of obesity-specific quality of life. IWQOL-Lite provides an overall total score as well as scores on five domains: (1) physical function, (2) self-esteem, (3) sexual life, (4) public distress, and (5) work. The raw scores will be transformed as follows (Tessier et al, 2012): the transformed scores range from 0 to 100, with 100 representing the best, and 0 representing the most impaired quality of life.

$$Transformed\ Score = \frac{maximum\ theoretical\ score - actual\ score}{test\ score\ range} X100$$

CGI-S response will be categorized into the categories summarized in Table 1. The number and percentage of subjects in each category and with shifts from baseline will be summarized based on the observed data by descriptive statistics at 1, 3, 6, and 12 months. The shift categories are summarized in Table 2.

**Table 1: Definition of Shift CGI-S Categories** 

| Response Category | CGI-S Score |
|---------------------------|-------------|
| Markedly to Extremely Ill | ≥5 |
| Moderately III | 4 |
| Normal to Mildly Ill | ≤3 |

#### **Table 2:** Shift Categories for CGI-S response

# Shift from Baseline Category for CGI-S Response Baseline Category Shift Category Markedly to Extremely Ill No change

2 level improvement

Moderately III
No change

1 level improvement

≥1 level improvement

1 level worsening

Normal to Mildly Ill

No change

≥1 level worsening

2 level worsening

Time to treatment discontinuation will be analyzed using the Kaplan-Meier method and the KM plot will be provided. Both all-cause discontinuation and discontinuation due to AE will be summarized. For prematurely discontinued subjects (all cause or due to AE), time to event is defined as time from the date of first dose of study drug in study ALK3831-A308 to the date of last dose of study drug. Other subjects will be censored at the last dose of the study drug.

#### 3.7.2. Multiple Comparison / Multiplicity

Not applicable.

#### 3.7.3. Subgroup Analysis

Subgroup analyses of efficacy endpoints will be performed for each of the following categories:

- Bipolar disorder
  - Change from baseline in IWQOL-Lite score by visit
  - Weight, metabolic responses, waist circumference, safety AEs and shift in CGI score in 2 points or 5 compared to those hospitalized due to AEs will be presented by visit.
- Sex (male, female)
- Age (<18 years,  $\ge 18$  years)
- Age (<30 years,  $\ge 30$  years)
- Race (Black or African American, Non-Black or Non-African American)

- Baseline BMI (<25 kg/m2,  $\ge 25 \text{ kg/m2}$ )
- Region (US, Non-US)
- Among those who completed study at 24 months, 36 months, and 48 months, change in weight, waist circumference and metabolic responses will be summarized.
- For those who switched from ALKS3831-A307 to ALKS3831-A308 change from baseline in CGI, weight, waist circumference and lipid levels by visit will be summarized.

Descriptive statistics will be provided for the subgroups listed above.

#### 3.7.4. Other Endpoints

Other endpoints include:

- Absolute change from baseline in fasting lipids (triglycerides, LDL, HDL, total cholesterol, fasting glucose, hemoglobin A1c (HbA1c), insulin) by subgroups
- Absolute change from baseline in fasting lipids (triglycerides, LDL, HDL, total cholesterol, fasting glucose, hemoglobin A1c (HbA1c), insulin) by antecedent study at End of the treatment
- Absolute change from baseline in BMI by visit
- BMI shift:
  - Proportion of subjects shifting from BMI <25 kg/m2 at baseline to BMI ≥25 kg/m2 by visit</li>
  - Proportion of subjects shifting from BMI <30 kg/m2 at baseline to BMI ≥30 by visit

### 3.8. Safety Analysis

All safety endpoints will be summarized for the Safety Population.

#### 3.8.1. Adverse Events

Incidence of treatment-emergent AEs (TEAEs) will be analyzed as a safety endpoint. Adverse events will be coded by System Organ Class and Preferred Term using the Medical Dictionary for Regulatory Activities (MedDRA®) Version 21.0 or higher. The verbatim term will be included in the AE listings.

An AE (coded by preferred term) will be considered a TEAE if the event is newly occurring or worsening on or after the date of first dose of study drug and within 7 days after the last dose of study drug in this study.

An overview table, including number of subjects with TEAEs, AEs leading to treatment discontinuation, study drug related TEAEs, and SAEs will be provided.

The number and percentage of subjects reporting TEAEs during the treatment period will be presented for the following categories:

- System organ class and preferred term
- Preferred term, and including the following subset:
  - TEAEs experienced by ≥2% of subjects
- System organ class, preferred term, and severity
- System organ class, preferred term for severe TEAEs
- System organ class, preferred term, and relationship
- System organ class, preferred term for study drug related TEAEs

If the same preferred term occurred more than once for the same subject, the subject will be counted only once for that preferred term using the most severe and most related occurrence for the summarization by severity and by relationship to the study drug.

In addition, the number and percentage of subjects reporting AEs during the safety follow-up period will be tabulated by the system organ class and preferred term.

Subgroup analysis by age (<40 years vs ≥40 years), sex (Female vs Male) and race (Black or African American, White, and Other) will be performed for TEAEs during the treatment period by preferred term.

#### 3.8.1.1. Deaths, Serious and Other Significant AEs

The number and percentage of subjects who have serious adverse events (SAE) and AEs leading to discontinuation from the treatment will be summarized by system organ class and preferred term. And the number and percentage of subjects reporting SAEs will be summarized by system organ class, preferred term, and relationship to study drug.

By-subject listings will be provided for SAEs, AEs leading to treatment discontinuation and AEs leading to death.

#### 3.8.1.2. **AEs of Special Interest**

In addition, incidence of a selected subset of relevant AEs in this class of drugs (eg, TEAE to evaluate potential of movement disorders, TEAE to evaluate potential of suicidal ideation and behavior, etc.) will be summarized by preferred term. The selection of AEs per subset will be based on the preferred terms from Standardized MedDRA queries (SMQs) or Customized MedDRA queries (CMQs).

#### 3.8.2. Clinical Laboratory Parameters

Laboratory parameters will be presented in conventional (ie, US) units. Only scheduled laboratory parameters will be included in the summaries, unless specified otherwise. All laboratory data, including those collected at unscheduled visits, will be included in the listings.

Laboratory results including baseline and change from baseline for the Safety Population during the treatment period for chemistry and hematology parameters will be summarized by visit.

Clinical laboratory test values, scheduled or unscheduled, will be considered potentially clinically significant (PCS) if they meet PCS criteria listed in Table 3. The number and

percentage of subjects who have postbaseline PCS clinical laboratory values will be summarized. The percentages will be calculated based on the number of subjects with abnormal baseline value and have at least one postbaseline assessment. All PCS values including baseline PCS values will be included in supportive listings.

Shift tables for selected fasting metabolic parameters (glucose, total cholesterol, low density lipoprotein [LDL], high density lipoprotein [HDL], triglycerides, and hemoglobin A1c [HbA1c]) and liver function tests will be presented. The criteria are summarized in Table 4, Table 5, and Table 6.

Table 3: Criteria of Potentially Clinically Significant (PCS) Abnormality for Selected Analytes

| Parameter Criteria | |
|-----------------------------------|-----------------------------|
| Chemistry | |
| Albumin | <2 g/dL |
| Alkaline Phosphatase (U/L) | ≥3 × ULN |
| Alanine Aminotransferase (U/L) | ≥3 × ULN |
| Aspartate Aminotransferase (U/L) | ≥3 × ULN |
| Bilirubin, Total | ≥2.0 mg/dL |
| Blood Urea Nitrogen | >30 mg/dL |
| Cholesterol, Random | >400 mg/dL |
| Cholesterol, Fasting <sup>a</sup> | ≥240 mg/dL |
| Cholesterol, Fasting | Increase ≥40 mg/dL |
| Cholesterol, HDL Fasting | <40 mg/dL |
| Cholesterol, HDL Fasting | Decrease ≥20 mg/dL |
| Cholesterol, LDL Fasting | ≥160 mg/dL |
| Cholesterol, LDL Fasting | Increase ≥30 mg/dL |
| Creatine Kinase (U/L) | ≥3 × ULN |
| Creatinine | ≥2.0 mg/dL |
| Glucose, Random | <40 mg/dL or<br>≥250 mg/dL |
| Glucose, Fasting | <50 mg/dL or<br>≥126 mg/dL |
| Glucose, Fasting | Increase ≥10 mg/dL |
| HbA1c | ≥5.7% |
| Potassium | <3 mmol/L or<br>>5.5 mmol/L |
| Lactate Dehydrogenase (U/L) | >3 × ULN |

| Parameter | Criteria |
|---|---|
| Prolactin (Female) | ≥ 1 X ULN <sup>b</sup> |
| Prolactin (Male) | ≥ 1 X ULN <sup>b</sup> |
| Prolactin (Female) | ≥ 3 X ULN <sup>b</sup> |
| Prolactin (Male) | ≥ 3 X ULN <sup>b</sup> |
| Sodium | <130 mmol/L or<br>>150 mmol/L |
| Triglycerides, Fasting | ≥200 mg/dL |
| Triglycerides, Fasting | Increase ≥50 mg/dL |
| Hematology | |
| Eosinophils | $>1.0 \times 10^3/\mu$ L |
| Hematocrit (Female) | ≤32% |
| Hematocrit (Male) | ≤37% |
| Neutrophils, Absolute | $<1.5\times10^3/\mu L$ |
| Platelets | $<75.0 \times 10^3 \text{ cells/}\mu\text{L or}$<br>$\geq 700.0 \times 10^3 \text{ cells/}\mu\text{L}$ |
| Leukocytes | $\leq 2.8 \times 10^{3}/\mu L \text{ or } \\ \geq 16.0 \times 10^{3}/\mu L$ |

<sup>&</sup>lt;sup>a</sup> Reported fasting

Table 4: Shifts Category from Baseline to Any Postbaseline for Selected Lipid Parameters

| Total Cholesterol (fasting) mg/dL |
|---------------------------------------------|
| Normal (<200) to High (≥240) |
| Borderline (≥200 and < 240) to High (≥240) |
| Normal (<200) to Borderline (≥200 and <240) |
| LDL Cholesterol (fasting) mg/dL |
| Normal (<100) to High (≥160) |
| Borderline (≥100 and <160) to High (≥160) |
| Normal (<100) to Borderline (≥100 and <160) |
| HDL Cholesterol (fasting) mg/dL |
| Normal (≥40) to Low (<40) |
| Triglycerides (fasting) mg/dL |
| Normal (<150) to High (≥200) |

<sup>&</sup>lt;sup>b</sup> ULN is 30 ng/mL for females and 20 ng/mL for males

| Borderline (≥150 and <200) to High (≥200) |
|---------------------------------------------|
| Normal (<150) to Borderline (≥150 and <200) |

#### Table 5: Shift Category from Baseline to Any Postbaseline in Glucose and HbA1c

| Glucose (fasting) mg/dL |
|------------------------------------------------|
| Normal (<100) to Impaired (≥100 and <126) |
| Normal (<100) to High (≥126) |
| Impaired (≥100 and <126) to High (≥126) |
| HbA1c % |
| Normal (<5.7%) to Borderline (≥5.7% and <6.5%) |
| Borderline (≥5.7% and <6.5%) to High (≥6.5%) |
| Normal (<5.7%) to High (≥6.5%) |

#### Table 6: Shift Category from Baseline to Any Postbaseline in Liver Function Test

| Alanine Aminotransferase (ALT) (U/L) |
|----------------------------------------|
| Shift from Normal to ≥3 x ULN |
| Shift from Normal to ≥5 x ULN |
| Shift from Normal to ≥10 x ULN |
| Aspartate Aminotransferase (AST) (U/L) |
| Shift from Normal to ≥3 x ULN |
| Shift from Normal to ≥5 x ULN |
| Shift from Normal to ≥10 x ULN |
| Bilirubin, Total (mg/dL) |
| Shift from Normal to >1 x ULN |
| Shift from Normal to ≥2 x ULN |

#### 3.8.3. Vital Signs and Body Weight

#### **3.8.3.1.** Vital Signs

Descriptive statistics for vital signs and changes from baseline values at each scheduled time point will be presented for the treatment period.

Vital sign values will be considered PCS if they meet both the observed-value criteria and the change-from-baseline criteria listed in Table 7. The number and percentage of subjects with PCS postbaseline values will be tabulated. The percentages will be calculated based on the number of subjects with abnormal baseline values and at least one postbaseline assessment. The numerator will be the number of subjects with abnormal baseline values and at least one postbaseline PCS value. A supportive listing of subjects with PCS postbaseline values will be provided.

All vital signs will be presented in the subject data listing.

Table 7: Criteria for Potentially Clinically Significant (PCS) Blood Pressure or Pulse Rate

| Parameter | Criteria |
|---|---|
| Supine Systolic Blood Pressure | ≤90 and decrease ≥20 mm Hg<br>≥180 and increase ≥20 mm Hg |
| Supine Diastolic Blood Pressure | ≤50 and decrease ≥15 mm Hg<br>≥105 and increase ≥15 mm Hg |
| Supine Heart Rate | ≤50 and decrease ≥15 bpm<br>≥120 and increase ≥15 bpm |

### 3.8.3.2. Weight and Body Mass Index

Weight (kg), BMI (kg/m²) and waist circumferences (cm) (baseline and change from baseline) will be summarized using observed data. Absolute and percent change from baseline in body weight will be summarized.

Number and percentage of subjects with  $\geq 7\%$  or  $\geq 10\%$  weight gain from baseline based on the observed data will be summarized by visit. Subgroup analysis by region (US vs non-US) will be performed. In addition, number and percentage of subjects with weight change values considered as PCS occurring at any post-baseline visit will be summarized. Criteria for PCS are presented below in Table 8. The percentages will be calculated relative to the number of subjects in the Safety Population with at least one post-baseline value. A supportive listing will be provided for subjects with PCS values.

Table 8: Criteria for Potentially Clinically Significant (PCS) Changes from Baseline in Body Weight

| Parameter | Criteria |
|-------------|----------------------------------------------------------|
| Body Weight | Decrease from Baseline ≥7%<br>Increase from Baseline ≥7% |

#### 3.8.4. Columbia-Suicide Severity Rating Scale (C-SSRS)

The C-SSRS is a questionnaire used to measure the presence and intensity of suicidal ideation and behavior (Table 9).

Suicidal behavior and suicidal ideation will be summarized for the Safety Population. The number of subjects with suicidal ideation and suicidal behavior will be summarized when applicable.

Supportive tabular display of subjects with all values will be provided.

**Table 9:** C-SSRS Categories for Analysis

| Category | C-SSRS Item response is "YES" |
|---|---|
| Suicidal behavior <sup>a</sup> | Preparatory acts or behavior |
| | Aborted attempt |
| | Interrupted attempt |
| | Actual attempt |
| | Complete suicide |
| Suicidal ideation <sup>a</sup> | Wish to be dead |
| | Non-specific active suicidal thoughts |
| | Active suicidal ideation with any methods (not plan) without intent to act |
| | Active suicidal ideation with some intent to act, without specific plan |
| | Active suicidal ideation with specific plan and intent |
| Non-Suicidal Self-Injurious | Non-Suicidal Self-Injurious |
| Behavior | Behavior |

<sup>&</sup>lt;sup>a</sup> Derived based on responses to individual items listed within the category

#### 3.9. Pharmacokinetic/ Pharmacodynamic Data Analysis

Not applicable.

#### 4. INTERIM ANALYSES

As described in Section 1, this SAP document is an update of the interim analysis that was conducted to support the ALKS 3831 New Drug Application (NDA). The full study population will be analyzed once the study is completed.

# 5. CHANGES IN CONDUCT OR PLANNED ANALYSES FROM THE PROTOCOL

To further assess the long-term durability, the following analysis was added in ISAP but was not specified in protocol:

• Shift analysis in CGI-S

# 6. DEFINITIONS AND CONVENTIONS FOR HANDLING OF THE DATA

Dataset specifications will be provided in a separate document.

### **6.1.** Analysis Visit Windows

Scheduled analysis visits are visits at scheduled timepoints as specified in the protocol (Table 1).

Scheduled analysis visits during the study period will be the same as the nominal visits collected in eCRF. There will be one valid value of assessment kept for each scheduled analysis visit in summary/analysis statistics.

Unscheduled visits are visits with data not collected on the scheduled time point. Unscheduled visits will not be used for by-visit summary/analysis statistics, unless specified otherwise.

All unscheduled visits as collected in eCRF will be included in listings.

Last postbaseline values are defined as the last valid postbaseline values collected for each subject during the treatment period.

An early termination (ET) visit during the on-treatment period can be mapped to a scheduled visit, if there is no valid value already at that visit. Visit window as defined in Table 10 for weight, waist circumference and CGI-S data and Table 11 for vital signs, lab and IWQOL-Lite data will be used to map the assessments collected after premature discontinuation of the study drug. An ET visit that is not mapped will not be summarized in the tables or figures but will be included in the listing.

Table 10: Visit Window Definition for Weight, Waist Circumference and CGI-S Data

| Analysis Visit to be<br>Mapped to | Target Study Month | Target Visit Date | Visit Window |
|---|---|---|---|
| Visit 2 | Month 1 | Day 29 | [2, 42] |
| Visit 3 | Month 2 | Day 57 | [43, 70] |
| Visit 4 | Month 3 | Day 85 | [71, 98] |
| Visit 5 | Month 4 | Day 113 | [99, 126] |
| Visit 6 | Month 5 | Day 141 | [127, 154] |
| Visit 7 | Month 6 | Day 169 | [155, 182] |
| Visit 8 | Month 7 | Day 197 | [183, 210] |
| Visit 9 | Month 8 | Day 225 | [211, 238] |
| Visit 10 | Month 9 | Day 253 | [239, 266] |
| Visit 11 | Month 10 | Day 281 | [267, 294] |
| Visit 12 | Month 11 | Day 309 | [295, 322] |
| Visit 13 | Month 12 | Day 337 | [323, 350] |
| Visit 14 | Month 13 | Day 365 | [351, 378] |
| Visit 15 | Month 14 | Day 393 | [379, 406] |
| Visit 16 | Month 15 | Day 421 | [407, 434] |
| Visit 17 | Month 16 | Day 449 | [435, 462] |

| Analysis Visit to be<br>Mapped to | Target Study Month | Target Visit Date | Visit Window |
|---|---|---|---|
| Visit 18 | Month 17 | Day 477 | [463, 490] |
| Visit 19 | Month 18 | Day 505 | [491, 518] |
| Visit 20 | Month 19 | Day 533 | [519, 546] |
| Visit 21 | Month 20 | Day 561 | [547, 574] |
| Visit 22 | Month 21 | Day 589 | [575, 602] |
| Visit 23 | Month 22 | Day 617 | [603, 630] |
| Visit 24 | Month 23 | Day 645 | [631, 658] |
| Visit 25 | Month 24 | Day 673 | [659, 686] |
| Visit 26 | Month 25 | Day 701 | [687, 714] |
| Visit 27 | Month 26 | Day 729 | [715, 742] |
| Visit 28 | Month 27 | Day 757 | [743, 770] |
| Visit 29 | Month 28 | Day 785 | [771, 798] |
| Visit 30 | Month 29 | Day 813 | [799, 826] |
| Visit 31 | Month 30 | Day 841 | [827, 854] |
| Visit 32 | Month 31 | Day 869 | [855, 882] |
| Visit 33 | Month 32 | Day 897 | [883, 910] |
| Visit 34 | Month 33 | Day 925 | [911, 938] |
| Visit 35 | Month 34 | Day 953 | [939, 966] |
| Visit 36 | Month 35 | Day 981 | [967, 994] |
| Visit 37 | Month 36 | Day 1009 | [995, 1022] |
| Visit 38 | Month 37 | Day 1037 | [1023, 1050] |
| Visit 39 | Month 38 | Day 1065 | [1051, 1078] |
| Visit 40 | Month 39 | Day 1093 | [1079, 1106] |
| Visit 41 | Month 40 | Day 1121 | [1107, 1134] |
| Visit 42 | Month 41 | Day 1149 | [1135, 1162] |
| Visit 43 | Month 42 | Day 1177 | [1163, 1190] |
| Visit 44 | Month 43 | Day 1205 | [1191, 1218] |
| Visit 45 | Month 44 | Day 1233 | [1219, 1246] |
| Visit 46 | Month 45 | Day 1261 | [1247, 1274] |
| Visit 47 | Month 46 | Day 1289 | [1275, 1302] |
| Visit 48 | Month 47 | Day 1317 | [1303, 1330] |

| Analysis Visit to be<br>Mapped to | Target Study Month | Target Visit Date | Visit Window |
|---|---|---|---|
| Visit 49 | Month 48 | Day 1345 | [1331, 1351] |

Visit Day is calculated as visit date – date of the first dose of study drug + 1. 1 month=28 days

Table 11: Visit Window Definition for Vital Signs, Lab and IWQOL-Lite Data

| Analysis Visit to be<br>Mapped to | Target Study Month | Target Visit Day | Visit Window |
|---|---|---|---|
| Visit 4 | Month 3 | Day 85 | [2, 126] |
| Visit 7 | Month 6 | Day 169 | [127, 210] |
| Visit 10 | Month 9 | Day 253 | [211, 294] |
| Visit 13 | Month 12 | Day 337 | [295, 378] |
| Visit 16 | Month 15 | Day 421 | [379, 462] |
| Visit 19 | Month 18 | Day 505 | [463, 546] |
| Visit 22 | Month 21 | Day 589 | [547,630] |
| Visit 25 | Month 24 | Day 673 | [631,714] |
| Visit 28 | Month 27 | Day 757 | [715,798] |
| Visit 31 | Month 30 | Day 841 | [799, 882] |
| Visit 34 | Month 33 | Day 925 | [883,966] |
| Visit 37 | Month 36 | Day 1009 | [967,1050] |
| Visit 40 | Month 39 | Day 1093 | [1051,1134] |
| Visit 43 | Month 42 | Day 1177 | [1135,1218] |
| Visit 46 | Month 45 | Day 1261 | [1219,1302] |
| Visit 49 | Month 48 | Day 1345 | [1303,1351] |

Visit Day is calculated as visit date – date of the first dose of study drug + 1. 1 month=28 days

# **6.2.** Handling of Partial Dates of Concomitant Medication and Adverse Events

Partial start dates of prior, concomitant medications, and adverse events will be assumed to be the earliest possible date consistent with the partial date. Partial stop dates of prior, concomitant medications, and adverse events will be assumed to be the latest possible date consistent with the partial date. In the case of completely missing stop date, medication will be assumed to be ongoing.

## 6.3. Handling of Safety Data

All efforts should be made to obtain the missing information from the investigator. For C-SSRS, vital signs and laboratory testing (chemistry, hematology, urinalysis), only observed data will be used for analyses, and missing data will not be imputed.

# 7. GENERAL STATISTICAL METHODOLOGY (AND REPORTING OF RESULTS)

In general, summary statistics (n, mean, SD, median, minimum, and maximum for continuous variables, and number and percentage of subjects in each category for categorical variables) will be provided. All summary tables will be based on observed data, and missing values will not be imputed, unless otherwise indicated. Measurements collected from unscheduled visits or repeated assessments will not be included in the by-visit summary tables or figures but will be included in the analyses for the PCS postbaseline values, and subject listings. Source data for the summary tables will be presented as subject data listings.

### 7.1. Reporting Precision

Summary statistics will be presented to the following degree of precision (Table 12), unless otherwise specified:

**Table 12:** Degree of Precision

| Statistics | Degree of Precision |
|---|---|
| Mean, Median, Confidence limit boundaries | One more than the raw data, up to 3 decimal places. |
| Standard deviation, Standard error | One more than the mean, up to 3 decimal places |
| Minimum, Maximum | The same as the raw data, up to 2 decimal places |
| P-value | Rounded to 3 decimal places and therefore presented as 0.xxx; <i>P</i> -values smaller than 0.001 as '<0.001'; P-values greater than 0.999 as '>0.999'. |
| Percentage | One decimal place. A percentage of 100% will be reported as 100%. Percentages of zero will be reported as 0. |

Fractional numeric values will be presented with a zero to the left of the decimal point (for example, 0.12 - 0.30).

For weight, height, and body mass index (BMI), one decimal place will be used for summary statistics, unless otherwise specified.

#### 8. PROGRAMMING SPECIFICATIONS

Programming specifications will be provided in a separate document.

# 9. MOCK TABLES, LISTINGS AND FIGURES (TLFS)

Mock-up tables and listings will be provided in a separate document.

# 10. REFERENCES

Tessier A, Zavorsky GS, Kim dJ, Carli F, Christou N, Mayo NE. Understanding the Determinants of Weight-Related Quality of Life among Bariatric Surgery Candidates. *J Obes*. 2012;2012:713426. doi: 10.1155/2012/713426.

# APPENDIX 1. AESI - MOVEMENT DISORDERS (INCLUDING EXTRAPYRAMIDAL SYNDROME AND TARDIVE DYSKINESIA; STANDARDIZED MEDDRA QUERY)

| Preferred Term (SMQ [#20000095] of Extrapyramidal syndrome) | PT Code |
|-------------------------------------------------------------|----------|
| Abnormal involuntary movement scale | 10075002 |
| Action tremor | 10072413 |
| Akathisia | 10001540 |
| Akinesia | 10001541 |
| Athetosis | 10003620 |
| Ballismus | 10058504 |
| Blepharospasm | 10005159 |
| Bradykinesia | 10006100 |
| Bradyphrenia | 10050012 |
| Buccoglossal syndrome | 10006532 |
| Chorea | 10008748 |
| Choreoathetosis | 10008754 |
| Chronic tic disorder | 10076661 |
| Cogwheel rigidity | 10009848 |
| Complex tic | 10076663 |
| Dopamine dysregulation syndrome | 10067468 |
| Drooling | 10013642 |
| Dyskinesia | 10013916 |
| Dyskinesia hyperpyrexia syndrome | 10071302 |
| Dyskinesia neonatal | 10013922 |
| Dyskinesia oesophageal | 10013924 |
| Dysphonia | 10013952 |
| Dystonia | 10013983 |
| Dystonic tremor | 10073210 |
| Emprosthotonus | 10014566 |
| Extrapyramidal disorder | 10015832 |
| Facial spasm | 10063006 |
| Fine motor skill dysfunction | 10076288 |
| Freezing phenomenon | 10060904 |

| Preferred Term (SMQ [#20000095] of Extrapyramidal syndrome) | PT Code |
|-------------------------------------------------------------|----------|
| Gait disturbance | 10017577 |
| Gait inability | 10017581 |
| Grimacing | 10061991 |
| Hyperkinesia | 10020651 |
| Hyperkinesia neonatal | 10020652 |
| Hypertonia | 10020852 |
| Hypertonia neonatal | 10048615 |
| Hypokinesia | 10021021 |
| Hypokinesia neonatal | 10021022 |
| Hypokinetic dysarthria | 10082243 |
| Laryngeal tremor | 10078751 |
| Laryngospasm | 10023891 |
| Meige's syndrome | 10027138 |
| Micrographia | 10057333 |
| Mobility decreased | 10048334 |
| Motor dysfunction | 10061296 |
| Movement disorder | 10028035 |
| Muscle contractions involuntary | 10028293 |
| Muscle rigidity | 10028330 |
| Muscle spasms | 10028334 |
| Muscle spasticity | 10028335 |
| Muscle tightness | 10049816 |
| Muscle tone disorder | 10072889 |
| Muscle twitching | 10028347 |
| Musculoskeletal stiffness | 10052904 |
| Oculogyric crisis | 10030071 |
| Oesophageal spasm | 10030184 |
| On and off phenomenon | 10030312 |
| Opisthotonus | 10030899 |
| Oromandibular dystonia | 10067954 |
| Oropharyngeal spasm | 10031111 |
| Parkinsonian crisis | 10048868 |

| Preferred Term (SMQ [#20000095] of Extrapyramidal syndrome) | PT Code |
|-------------------------------------------------------------|----------|
| Parkinsonian gait | 10056242 |
| Parkinsonian rest tremor | 10056437 |
| Parkinsonism | 10034010 |
| Parkinsonism hyperpyrexia syndrome | 10071243 |
| Parkinson's disease | 10061536 |
| Parkinson's disease psychosis | 10074835 |
| Pharyngeal dyskinesia | 10070912 |
| Pharyngeal dystonia | 10081226 |
| Pleurothotonus | 10035628 |
| Postural reflex impairment | 10067206 |
| Postural tremor | 10073211 |
| Posture abnormal | 10036436 |
| Posturing | 10036437 |
| Propulsive gait | 10082328 |
| Protrusion tongue | 10037076 |
| Provisional tic disorder | 10076694 |
| Psychomotor hyperactivity | 10037211 |
| Rabbit syndrome | 10068395 |
| Reduced facial expression | 10078576 |
| Respiratory dyskinesia | 10057570 |
| Resting tremor | 10071390 |
| Restlessness | 10038743 |
| Risus sardonicus | 10039198 |
| Secondary tic | 10076702 |
| Spasmodic dysphonia | 10067672 |
| Status dystonicus | 10088053 |
| Tardive dyskinesia | 10043118 |
| Tic | 10043833 |
| Tongue spasm | 10043981 |
| Torticollis | 10044074 |
| Torticollis psychogenic | 10044076 |
| Tremor | 10044565 |

| Preferred Term (SMQ [#20000095] of Extrapyramidal syndrome) | PT Code |
|-------------------------------------------------------------|----------|
| Tremor neonatal | 10044575 |
| Trismus | 10044684 |
| Uvular spasm | 10050908 |
| Walking disability | 10053204 |
| Writer's cramp | 10072249 |

# APPENDIX 2. AESI - SUICIDAL IDEATION AND BEHAVIOR (CUSTOM MedDRA QUERY)

| Preferred Term | PT Code |
|-------------------------------------------------|----------|
| Assisted suicide | 10079105 |
| Columbia suicide severity rating scale abnormal | 10075616 |
| Completed suicide | 10010144 |
| Depression suicidal | 10012397 |
| Intentional overdose | 10022523 |
| Intentional self-injury | 10022524 |
| Overdose | 10033295 |
| Poisoning deliberate | 10036000 |
| Self-injurious ideation | 10051154 |
| Suicidal behaviour | 10065604 |
| Suicidal ideation | 10042458 |
| Suicide attempt | 10042464 |
| Suicide threat | 10077417 |
| Suspected suicide | 10082458 |
| Suspected suicide attempt | 10081704 |

# APPENDIX 3. AE TERMS - ABUSE POTENTIAL (CUSTOM MedDRA QUERY)

| Category | Preferred Term | PT Code |
|----------------|-----------------------------------------------|----------|
| Abuse behavior | Accidental overdose | 10000381 |
| | Drug abuse | 10013654 |
| | Drug abuser | 10061111 |
| | Drug detoxification | 10052237 |
| | Drug diversion | 10066053 |
| | Drug level above therapeutic | 10061132 |
| | Drug level increased | 10013722 |
| | Drug screen | 10050837 |
| | Drug screen positive | 10049177 |
| | Drug use disorder | 10079381 |
| | Drug use disorder, antepartum | 10079382 |
| | Drug use disorder, postpartum | 10079383 |
| | Intentional overdose | 10022523 |
| | Intentional product misuse | 10074903 |
| | Intentional product use issue | 10076308 |
| | Maternal use of illicit drugs | 10026938 |
| | Needle track marks | 10028896 |
| | Neonatal complications of substance abuse | 10061862 |
| | Overdose | 10033295 |
| | Prescription drug used without a prescription | 10076639 |
| | Prescription form tampering | 10067669 |
| | Product tampering | 10069330 |
| | Reversal of opiate activity | 10039004 |
| | Substance abuse | 10066169 |
| | Substance abuser | 10067688 |
| | Substance use | 10070964 |
| | Substance use disorder | 10079384 |
| | Substance-induced mood disorder | 10072387 |
| | Substance-induced psychotic disorder | 10072388 |
| | Toxicity to various agents | 10070863 |

| Category | Preferred Term | PT Code |
|------------------|------------------------------------------|----------|
| Euphoria related | Euphoric mood | 10015535 |
| | Feeling abnormal | 10016322 |
| | Feeling drunk | 10016330 |
| | Feeling of relaxation | 10016352 |
| | Hallucination | 10019063 |
| | Hallucination, auditory | 10019070 |
| | Hallucination, gustatory | 10019071 |
| | Hallucination, olfactory | 10019072 |
| | Hallucination, synaesthetic | 10062824 |
| | Hallucination, tactile | 10019074 |
| | Hallucination, visual | 10019075 |
| | Hallucinations, mixed | 10019079 |
| | Inappropriate affect | 10021588 |
| | Mood altered | 10027940 |
| | Mood swings | 10027951 |
| | Thinking abnormal | 10043431 |
| Non-specific | Acute psychosis | 10001022 |
| | Aggression | 10001488 |
| | Cognitive disorder | 10057668 |
| | Confusional state | 10010305 |
| | Delirium | 10012218 |
| | Delusional disorder, unspecified type | 10012255 |
| | Depersonalisation/derealisation disorder | 10077805 |
| | Disorientation | 10013395 |
| | Dissociation | 10013457 |
| | Disturbance in attention | 10013496 |
| | Disturbance in social behaviour | 10061108 |
| | Dopamine dysregulation syndrome | 10067468 |
| | Emotional disorder | 10014551 |
| | Flight of ideas | 10016777 |
| | Medication overuse headache | 10072720 |

| Category | Preferred Term | PT Code |
|----------|-------------------------|----------|
| | Mental impairment | 10027374 |
| | Narcotic bowel syndrome | 10072286 |
| | Paranoia | 10033864 |
| | Psychotic behaviour | 10037249 |
| | Psychotic disorder | 10061920 |
| | Sedation | 10039897 |
| | Stupor | 10042264 |

# APPENDIX 4. AE TERMS – DEPENDENCE (CUSTOM MedDRA QUERY)

| Preferred Term | PT Code |
|-----------------------------|----------|
| Dependence | 10012335 |
| Drug dependence | 10013663 |
| Drug dependence, antepartum | 10013675 |
| Drug dependence, postpartum | 10013676 |
| Drug tolerance | 10052804 |
| Drug tolerance decreased | 10052805 |
| Drug tolerance increased | 10052806 |
| Substance dependence | 10076595 |

# APPENDIX 5. AE TERMS – WITHDRAWAL (CUSTOM MedDRA QUERY)

| Preferred Term | PT Code |
|-------------------------------------|----------|
| Abdominal pain | 10000081 |
| Agitation | 10001497 |
| Anhedonia | 10002511 |
| Anxiety | 10002855 |
| Arthralgia | 10003239 |
| Chills | 10008531 |
| Depressed mood | 10012374 |
| Depression | 10012378 |
| Diarrhoea | 10012735 |
| Drug detoxification | 10052237 |
| Drug rehabilitation | 10064773 |
| Drug withdrawal convulsions | 10013752 |
| Drug withdrawal headache | 10013753 |
| Drug withdrawal maintenance therapy | 10052970 |
| Drug withdrawal syndrome | 10013754 |
| Drug withdrawal syndrome neonatal | 10013756 |
| Dysphoria | 10013954 |
| Dyssomnia | 10061827 |
| Feeling of despair | 10016344 |
| Headache | 10019211 |
| Hyperhidrosis | 10020642 |
| Insomnia | 10022437 |
| Irritability | 10022998 |
| Morose | 10027977 |
| Mydriasis | 10028521 |
| Nausea | 10028813 |
| Negative thoughts | 10058672 |
| Nervousness | 10029216 |
| Obsessive thoughts | 10029897 |
| Pain | 10033371 |

| Preferred Term | PT Code |
|--------------------------------|----------|
| Persistent depressive disorder | 10077804 |
| Piloerection | 10035039 |
| Poor quality sleep | 10062519 |
| Rebound effect | 10038001 |
| Restlessness | 10038743 |
| Reversal of opiate activity | 10039004 |
| Rhinorrhoea | 10039101 |
| Steroid withdrawal syndrome | 10042028 |
| Syncope | 10042772 |
| Tachycardia | 10043071 |
| Terminal insomnia | 10068932 |
| Tremor | 10044565 |
| Vomiting | 10047700 |
| Withdrawal arrhythmia | 10047997 |
| Withdrawal syndrome | 10048010 |
| Yawning | 10048232 |

#### APPENDIX 6. COVID-19 ANALYSIS

Pandemic has resulted in certain disruptions in the study conduct since early 2020, including site closure, delayed study drug supply, subjects discontinuation and missing assessments. These impacts were limited in scope upon review of the protocol deviations, and also confounded by the initiation of new regions. Sites in Ukraine and Russia were first initiated in March 2020 and July 2020. Therefore, only descriptive statistics will be provided to explore the potential impact of the pandemic on the primary and secondary objectives of the study. The following subgroup analysis (before vs during pandemic) will be conducted:

- Disposition
- Demographics and Baseline Characteristics
- Protocol Deviation
- Primary Efficacy Endpoint
- Key Secondary Endpoints
- TEAE
- SAE

Subjects enrolled before 01 Mar 2020 will be grouped as before pandemic, and subjects enrolled after this date will be grouped as during pandemic. While the pandemic has started in various regions a few weeks apart, a single cutoff date will be applied.

# Signature Page for CLIN\_ALK3831-A308-sap

| Approved | Name: PPD<br>Capacity: Other<br>Date: 04-Dec-2023 19:59:22 GMT+0000 |
|---|---|
| Approved | Name: PPD<br>Capacity: Clinical<br>Date: 04-Dec-2023 23:33:04 GMT+0000 |
| Approved | Name: PPD Capacity: Clinical Date: 07-Dec-2023 12:34:29 GMT+0000 |
| Approved | Name: PPD Capacity: Other Date: 07-Dec-2023 13:00:52 GMT+0000 |

Alkermes® Confidential Information
Document REG-026019